CLINICAL TRIAL: NCT00128050
Title: Efficacy and Safety of Factor VIIa (Eptacog Alfa) on Rebleeding After Surgery for Spontaneous Supratentorial Intracerebral Hemorrhage. A Randomized, Controlled, Open-Label, Investigator-Blinded Pilot Study
Brief Title: Efficacy and Safety of Factor VIIa on Rebleeding After Surgery for Spontaneous Intracerebral Hemorrhage (ICH)
Acronym: PRE-SICH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Roberto Imberti, M.D., Fondazione IRCCS Policlinico S. Matteo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NS-SICH-2005
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Intracerebral Hemorrhage
Keywords: Spontaneous intracerebral hemorrhage; ICH; intracerebral rebleeding; cerebral hematoma evacuation; cerebral hematoma volume
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — recombinant FVIIa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients treated with recombinant FVIIa
  Interventions: Drug: rFactor VIIa (Eptacog alfa, NovoNordisk); Drug: rFVIIa
- 2 (Placebo Comparator): Patients with spontaneous supratentorial ICH included in this arm will be treated with placebo
  Interventions: Other: Sodiun chloride 0.9%

INTERVENTIONS:
Drug: rFactor VIIa (Eptacog alfa, NovoNordisk) — rFVIIa will be admistered as single bolus at the dosage of 100 mcg/Kg b.w.
  Arms: 1
Drug: rFVIIa — Patients with spontaneous supratentorial ICH will be treated with rFVII after hematoma evacuation
  Arms: 1
Other: Sodiun chloride 0.9% — Bolus injection of sodium chloride 0.9% after surgical hematoma removal
  Arms: 2

SUMMARY:
Although the role of surgical treatment is still controversial, surgical evacuation of intracerebral hematoma is a frequent practice. Rebleeding is a frequent complication in patients submitted to hematoma evacuation. It has been reported that smaller postoperative volume of hematoma is associated with a better outcome. The investigators hypothesize that the administration of Factor VIIa (Eptacog alfa) immediately after surgical evacuation of the hematoma can reduce postoperative rebleeding.

Aims of the Study:

This study will investigate:

1. The efficacy of Eptacog alfa in preventing or reducing rebleeding after surgery for spontaneous supratentorial ICH; and
2. The safety of product administration

DETAILED DESCRIPTION:
The primary endpoint is the evaluation of efficacy of Factor VIIa (Eptacog alfa, NovoSeven, Novo Nordisk) on rebleeding after surgery for primary supratentorial ICH. All patients included in the study will perform a CT scan within 3 hours before surgery, then immediately after surgery, and 18-30 hours after surgery. The hematoma volume will be evaluated by a multi-slice CT scan. All CT scan images will be sent to the Coordinating Center where the hematoma volume will be evaluated by a dedicated software by the same investigator who will be unaware of the treatment (investigator- blinded study).

SAFETY EVALUATION:

Seventeen episodes of thrombotic spontaneous adverse events have been reported after administration of 480,000 standard doses of Eptacog alfa in hemophilic patients. These episodes include myocardial infarction, acute cerebrovascular thrombosis, disseminated intravascular coagulation (DIC), deep venous thrombosis (DVT) and pulmonary embolism.

Before and after hematoma removal will be evaluated ECG, myocardiac enzymes, coagulation profile, CT scan (looking for ischemic events) and venous echodoppler ultrasound of lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years inclusive
* Intraparenchymal primary supratentorial intracerebral hemorrhage requiring surgical evacuation
* Any Glasgow Coma Score (GCS) score
* Surgery expected to be performed within 24 hours from symptoms onset

Exclusion Criteria:

* Age below 18
* Intraparenchymal hematoma secondary to rupture of cerebral aneurysm or bleeding of arteriovenous (A-V) malformation or cerebral tumors
* Contemporary involvement in another study
* Pregnancy
* Myocardial infarction in the six months preceding enrolment
* Coronary or carotid stents positioned in the six months preceding enrolment
* Solid organ transplant patients (e.g., heart, lung, liver, kidney)
* Pregnancy
* Myocardial infarction in the six months preceding enrolment
* Coronary and carotid stents positioned in the six months preceding enrolment
* Solid organ transplant patients (e.g., heart, lung, liver, kidney)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of Factor VIIa (Eptacog alfa) in preventing or reducing rebleeding after surgery for spontaneous supratentorial ICH | 4 years

SECONDARY OUTCOMES:
Safety of product administration | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Imberti, M.D., Principal Investigator — IRCCS Policlinico S. Matteo - Pavia - Italy
Locations (3):
- Italy (3):
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, Cuneo
  - Azienda Ospedaliera "Maggiore della Carità", Novara
  - II Dpt Anesthesiology&Critical Care Medicine - IRCCS Policlinico S. Matteo, Pavia

REFERENCES:
- [Background] Morgenstern LB, Demchuk AM, Kim DH, Frankowski RF, Grotta JC. Rebleeding leads to poor outcome in ultra-early craniotomy for intracerebral hemorrhage. Neurology. 2001 May 22;56(10):1294-9. doi: 10.1212/wnl.56.10.1294. PMID 11376176
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112